CLINICAL TRIAL: NCT01471314
Title: Functional MRI and MR Angiography Used in Spontaneous Migraine
Brief Title: MRA/fMRI Study of Spontaneous Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Faisal Mohammad Amin, MD, PhD student, Glostrup University Hospital, Copenhagen
Other Study IDs: H-C-2008-089
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Headache Versus Non-headache Day

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Spontaneous migraine
  Interventions: Behavioral: Headache day versus non-headache day

INTERVENTIONS:
Behavioral: Headache day versus non-headache day

SUMMARY:
The purpose of this study is to examine migraineurs during spontaneous migraine attacks without aura, using high resolution magnetic resonance imaging (MRI), to study following:

* Changes in resting state blood-oxygenation-level-dependent-signal (BOLD-signal) using functional MRI (fMRI).
* Changes in circumferences of intra- and extracranial arteries using MR-angiography (MRA).
* Changes in regional and global cerebral blood flow (CBF) using the arterial spin labeling (ASL) method.

Moreover to perform diffusion tensor imaging (DTI) scans during spontaneous migraine attacks.

The migraine specific drug sumatriptan will be given to relieve pain and the effect will be registered using MRA and fMRI if possible.

ELIGIBILITY:
Inclusion Criteria:

* Migraine without aura according to IHS criteria.

Exclusion Criteria:

* Other primary headaches.
* Tension-type headache more than 5 days/month.
* Use of anti-pain medication before the scanning on the examination day.
* Pregnant or nursing women.
* Contraindication for MR scan.
* Anamnestic or clinical signs of cardiovascular or cerebrovascular disease, unregulated psychiatric disease or drug misuse.
* Other clinical conditions assessed by the examining doctor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Migraine without aura
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup Hospital, Faculty of Health Sciences, University of Copenhagen, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Amin FM, Asghar MS, Hougaard A, Hansen AE, Larsen VA, de Koning PJ, Larsson HB, Olesen J, Ashina M. Magnetic resonance angiography of intracranial and extracranial arteries in patients with spontaneous migraine without aura: a cross-sectional study. Lancet Neurol. 2013 May;12(5):454-61. doi: 10.1016/S1474-4422(13)70067-X. Epub 2013 Apr 9. PMID 23578775